CLINICAL TRIAL: NCT02490462
Title: Impact of Physical Therapy Associated With a Program of Education of Caregivers in Functioning and Quality of Life of Children With Cerebral Palsy
Brief Title: Impact of an Education Program for Parents of Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Mansueto Gomes Neto, Mansueto Gomes Neto, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUBahia060278
Record Dates: First submitted 2015-05-06; First posted 2015-07-03 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Physical Therapy; Family-centered Care
MeSH Terms: conditions — Cerebral Palsy | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education + Conventional PhysicalTherapy (Experimental): Parents of children with cerebral palsy receive instructions for active inclusion of children in everyday activities. The education program for parents will take place once a week for twelve weeks. Children with Cerebral Palsy make conventional physical therapy twice a week for a period of twelve weeks.
  Interventions: Other: Education + Conventional PhysicalTherapy
- Conventional Physical Therapy (Active Comparator): Children with Cerebral Palsy make conventional physical therapy twice a week for a period of twelve weeks.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Education + Conventional PhysicalTherapy — The education program for parents will be held one day a week for 1 hour, with total duration of 12 weeks. During the parents or legal guardian meetings will be oriented to stimulate the drive to your child or ward during everyday activities such as bathing, dressing, eating, transferring, going to the bathroom. Parents will receive a diary to record the activities in the home environment. The orientation day for parents will take place in different days of the day the child will receive physical therapy, so that the physiotherapist responsible for the training of parents is shrouded in relation to the randomization of the subjects. This program will be associated with conventional physical therapy program that provides for movements based on neurodevelopmental concept.
  Arms: Education + Conventional PhysicalTherapy
Other: Conventional Physical Therapy — The full program will be for 24 weeks, the first step will consist of 12 weeks of training with a frequency of twice a week should total at least 18 Conventional physical therapy interventions and 09 meetings of guidelines for parents. After this step be performed to start new reviews second step further 12 weeks with the same characteristics as the first 12 weeks. The conventional physiotherapy program will consist of functional muscle training focused on the task. Tasks will be individualized based on the results of the evaluations of Gross Motor Function and Inventory Pediatric Evaluation of Disability. The sessions will last 45 minutes carried out 2 times a week, training will have a total duration of 12 weeks.
  Arms: Conventional Physical Therapy

SUMMARY:
The Physical Therapy for children with Cerebral Palsy is of great complexity, in addition to improving the neuromotor components at the level of structure and body function, must empower them to carry out their activities and daily tasks and enable their social participation. In this way, the goals of Physical Therapy are related to promote the independence and functionality of the individual in situations of daily life. The participation of caregivers in the rehabilitation process can contribute to potentiate the gains obtained by physical therapy as well as to which they are incorporated into the day to day management of children with cerebral palsy. Objective: To assess whether Physical Therapy associated with the education of caregivers is effective in improving the functioning and quality of life of children with cerebral palsy. Hypothesis: The combination of Physical therapy with the education of caregivers improves in 15% the parameters analyzed against only 10% in those who are only Physical Therapy. Methods: 60 children with cerebral palsy after acceptance and signature in the term of informed consent will be randomly divided into 2 groups (G1: Physiotherapy and education of caregivers and G2: only Physical Therapy) to do 3 sessions of Physical Therapy and 1 weekly session of group education with duration of 45 min during 12 consecutive weeks. The evaluation will be carried out by means of the System of Classification of Motor Function Gross (GMFCS), the evaluation of Motor Function through the scale GMFM-88 (Gross Motor Function Measure - 88 ) and the Activity and Participation will be evaluated by the Inventory of Evaluation of Pediatric Disability (PEDI). The analysis of the results will be carried out using the Statistical Package for the Social Sciences (SPSS) using descriptive statistics for social and demographic characteristics and inferential for normality of data (test Kolmogorov-Smirnov ), mean comparison test to check for differences between the groups and measures of association through the coefficient of correlation. The level of significance of 5% will be established

DETAILED DESCRIPTION:
Randomized clinical trial (RCT) in accordance with the recommendations of the Report of Consolidated Standards Trials (CONSORT) held in Clinical School of Physical Therapy, Federal University of Bahia (UFBA), Salvador, Bahia, with cerebral palsy patients and their caregivers. Selection of the population: Inclusion criteria 's own diagnosis of cerebral palsy for children, children will be included presenting grade I, II, III, IV and V in the System Gross Motor Function Classification (GMFCS) aged 1 year to 12 years old, and a parent or caregiver who dedicate themselves in full-time child, comply with the intervention protocol and sign the free and informed consent (IC). They will be deleted: Patients will be excluded disease of the peripheral nervous system or brain stem, children with other chronic diseases receiving palliative care, and children who have bone deformities such as scoliosis structured Cobb > 30 and lower limb deformity. A sample of 20 patients group is required. The sample size for the study was calculated, considering a statistical power of 80% to 5% alpha. Evaluation procedures: To measurement of motor function were used the Gross Motor Function Measure (GMFM-88) scales . The range consists of 5 sizes and each size is an engine development phase that is related to the first quarters of life. The GMFM-88 with respect to motor development stage presented by the child and the evaluator should assess only the dimensions that represent the stages of engine development for age. To check the Activity and Participation will be used Inventory Pediatric Disability Assessment (ASK). applied in children from 6 months to 7.5 years. It can also be used with older children who have functional limitations with performance below the expected for their age compared to typical children of the normative sample and can be used with children with various types of disabilities.

The ASK can be applied by any member of the interdisciplinary team through interviews with the caretaker. Each item is a task and the ability to realize it is scored as (1) whether the child is able and (0) if it is not able to perform it. Evaluates functional abilities and their performance in the areas of self-care (73 items), mobility (59 items) and social function (65 items).

Measures also the amount of assistance given by the caregiver when performing these tasks and the possible use of adaptations and changes in the environment. In caregiver assistance area for self-care are 8 items, 7 items mobility and social function 5 items. The score ranges from 0 to 5 (total dependence to complete independence).

To investigate the Quality of Life will use the Child Health Questionnaire (CHQ - PF50), in its version for parents, applicable to children through fifteen in health. Each concept has a score of 0-100, with higher scores indicating better health status, satisfaction and well-being, and result in two summary scores - physical and psychosocial (0-70). This questionnaire has been validated for children with cerebral palsy. All these measures will be evaluated in the pre-intervention, 4 weeks, 8 weeks and 12 weeks after initiation of therapy.

Procedure: Using Education will be a protocol for caregivers of children with cerebral palsy for the intervention group, once a week, while children in the control and intervention groups will receive conventional physical therapy twice a week. The established training period will last twelve weeks. Software to create randomization lists (randList®) is used in order to ensure that all individuals have equal chances allocation in groups.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral Palsy diagnosis for children,
2. Children will be included presenting grade II, III on Classification System of Gross Motor Function (GMFCS) aged 6 months to 12 years old.
3. Parent or caregiver who devote yourself full-time to the child,
4. Acceptance of parents for children to participate in the protocol by signing the free and informed consent form.

Exclusion Criteria:

1. Peripheral nervous system disease or brain stem
2. Children with other chronic diseases receiving palliative care,
3. Children who present bone deformity and scoliosis structured Cobb > 30 and lower limb deformity.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Functionality | 12 weeks
  Assess whether the associated physical therapy education of caregivers is effective in improving the functionality of children with cerebral palsy after a 12-week period.

SECONDARY OUTCOMES:
Gross Motor Function | 12 weeks
  To investigate the change in the gross motor function of children with cerebral palsy after physiotherapy intervention associated with an education program for parents.
  To measurement of motor function were used the GMFM-88 scales (Gross Motor Function Measure). The scales will be implemented before the start of the intervention and after six months of physiotherapy. The GMFM-88 consists of 88 items organized in five dimensions, the first lying and rolling, Sitting, crawling and Kneeling, Standing, Walking , Running and Jumping . The items are sorted within each dimension according to the practicality of execution within the overall assessment and difficulty. For each item, 0-3 notes are set, and the value 0 corresponds to the inactivity of the child in the requested activity.
Improvement in Functionality | 12 weeks
  Describe the functional profile of children with cerebral palsy according to the International Classification of Functioning.
  To check the Activity and Participation will be used Inventory Pediatric Disability Assessment (ASK). This review (25) is designed to be applied to children 6 months old to 7.5 years. It can also be used with older children who have functional limitations with performance below the expected for their age compared to typical children of the normative sample and can be used with children with various types of disabilities.
  The ASK can be applied by any member of the interdisciplinary team through interviews with the caretaker. Each item is a task and the ability to realize it is scored as (1) whether the child is able and (0) if it is not able to perform it. Evaluates functional abilities and their performance in the areas of self-care (73 items), mobility (59 items) and social function (65 items).
Motor performance and functional | 12 weeks
  To estimate the correlation engine and functional performance in children with cerebral palsy. It will be used the correlation test of Pearson or Spearman depending on the normality of the data, with information regarding the motor function and functionality.
Frequency of exercises | 12 weeks
  To investigate the influence of the regularity of carrying out household activities on the Gross Motor Function, Activity and Participation and Quality of life in children with cerebral palsy through a daily exercise.
  To assess the frequency of carrying out the activities, parents will receive a weekly diary with daily activities arranged in rows and days and shifts the willing week column. Should mark the days and corresponding shifts stimulation that performed in each functional activity.

CONTACTS AND LOCATIONS:
Overall Officials: Manseuto Gomes Neto, Principal Investigator — Federal University of Bahia
Locations (1):
- Mansueto Gomes Neto, Salvador, Estado de Bahia, Brazil